CLINICAL TRIAL: NCT05107375
Title: Clinical Study on Immunogenicity and Safety of Recombinant Novel Coronavirus（COVID-19）Vaccine (CHO Cell) Combined With Tetravalent Influenza Virus Lysis Vaccine in People Aged 18 Years and Over
Brief Title: Clinical Study of Recombinant Novel Coronavirus（COVID-19） Vaccine (CHO Cell) Combined With Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT-LKM-2021-NCV01
Record Dates: First submitted 2021-11-01; First posted 2021-11-04 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Coronavirus Disease 2019
Keywords: Recombinant Novel Coronavirus Vaccine; Tetravalent influenza virus lysis vaccine
MeSH Terms: conditions — COVID-19 | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population Ⅰ (Experimental): One dose of influenza virus split vaccine and one dose of recombinant Novel coronavirus vaccine (CHO cells) were given in the contralateral arm on day 0, the second dose of recombinant Novel coronavirus vaccine (CHO cells) on day 30 and the third dose of recombinant Novel coronavirus vaccine (CHO cells) on day 60, all in the upper arm deltoid muscle.
  Interventions: Biological: Tetravalent influenza virus lysis vaccine; Biological: Recombinant new coronavirus vaccine (CHO cell) group
- Population Ⅱ (Experimental): The first dose of recombinant Novel Coronavirus vaccine (CHO cells) was given on day 0, the second dose of recombinant Coronavirus vaccine (CHO cells) on day 30, the first dose of influenza virus lysate vaccine on day 44, and the third dose of recombinant Coronavirus vaccine (CHO cells) on day 60, all in the upper arm deltoid muscle.
  Interventions: Biological: Tetravalent influenza virus lysis vaccine; Biological: Recombinant new coronavirus vaccine (CHO cell) group

INTERVENTIONS:
Biological: Tetravalent influenza virus lysis vaccine — Influenza virus lysis vaccine, one dose at a time, each dose 0.5mL, containing each influenza virus strain hemagglutinin 15μg.
Biological: Recombinant new coronavirus vaccine (CHO cell) group — One dose of recombinant Novel Coronavirus vaccine (CHO cells) was administered at 0.5mL each dose, containing 25μg nCP-RBD protein.

SUMMARY:
Popular topic：Clinical study of recombinant Novel Coronavirus vaccine (CHO cell) combined with influenza vaccine. Research purpose:Main purpose:To evaluate the immunogenicity of recombinant Novel Coronavirus vaccine (CHO cells) combined with influenza vaccine in people aged 18 years and over. Secondary purpose:To evaluate the safety of recombinant Novel Coronavirus vaccine (CHO cells) combined with influenza vaccine in people aged 18 years and over. Overall design:An open experimental design was adopted in this study, and 300 subjects were planned to be enrolled. To evaluate the immunogenicity and safety of recombinant Novel Coronavirus vaccine (CHO cells) in combination with influenza vaccine. Study population:The study involved people 18 years of age and older.

Test groups:A total of 300 cases were enrolled. 240 patients in 18-59 years old group, 60 patients in ≥60 years old group. There were 150 cases in group A, 120 cases in 18-59 years old group, and 30 cases in ≥60 years old group. There were 150 cases in group B, 120 cases in 18-59 years old group and 30 cases in ≥60 years old group.

DETAILED DESCRIPTION:
Overall design:An open experimental design was adopted in this study, and 300 subjects were planned to be enrolled. To evaluate the immunogenicity and safety of recombinant Novel Coronavirus vaccine (CHO cells) in combination with influenza vaccine.

Intervention:

Group A: one dose of influenza virus split vaccine and one dose of recombinant Novel coronavirus vaccine (CHO cells) in the contralateral arm on day 0, the second dose of recombinant Novel coronavirus vaccine (CHO cells) on day 30, and the third dose of recombinant Novel coronavirus vaccine (CHO cells) on day 60 were given intramuscularly in the upper arm deltoid muscle.

Group B: the first dose of recombinant Novel coronavirus vaccine (CHO cells) was administered on day 0, the second dose of recombinant Coronavirus vaccine (CHO cells) on day 30, the first dose of influenza virus lysate vaccine on day 44, and the third dose of recombinant Coronavirus vaccine (CHO cells) on day 60.

One dose of recombinant Novel Coronavirus vaccine (CHO cells) was administered at 0.5mL each dose, containing 25μg nCP-RBD protein. Influenza virus lysis vaccine, one dose at a time, each dose 0.5mL, containing each influenza virus strain hemagglutinin 15μg.

Immunogenicity observation:

Evaluation of immunogenicity In group A, about 5.0mL of venous blood was collected for immunogenicity test before the first dose of vaccine, before the second dose of Novel Coronavirus vaccine (CHO cells) and 14 days after the third dose of recombinant Novel Coronavirus vaccine (CHO cells).

In group B, about 5.0mL of venous blood was collected for immunogenicity test before the first dose of vaccine and 14 days after the third dose of recombinant Novel Coronavirus vaccine (CHO cells).

Safety assessment

AE and SAE

All adverse events (AE), all AE at 30 min after each dose of recombinant Novel Coronavirus vaccine (CHO cells) and influenza vaccine, all AE at 0-7 days (both solicitation and non-solicitation AE) and all AE at 8-30 days (non-solicitation AE) were collected; All SAE were collected from the first dose to 1 month after full immunization.

Solicitation AE[the following events occurring within 7 days after vaccination with recombinant Novel Coronavirus vaccine (CHO cells)] :

Inoculation site (local) AE: pain, swelling, induration, redness, rash, pruritus Vital signs: fever Non-inoculated site (whole body) AE: headache, fatigue/fatigue, diarrhea, nausea, vomiting, muscle pain (non-inoculated site), acute allergic reaction, cough

Vital signs and physical examination

All subjects shall have their axillary body temperature checked daily during the screening period, before the subsequent dose of recombinant Novel Coronavirus vaccine (CHO cells), and within 7 days after each dose of recombinant Novel Coronavirus vaccine (CHO cells); Subjects in group B will have their armpit temperature measured before influenza vaccination (the day of vaccination).

All subjects underwent physical examination (skin and cardiopulmonary auscultation) and blood pressure measurement during the screening period.

Pregnancy event

Urine pregnancy test should be performed on women of childbearing age before each dose of recombinant Novel Coronavirus vaccine (CHO cells); Women of childbearing age in group B should have a urine pregnancy test prior to influenza vaccination.

Pregnancy events occurring within 1 month from the first dose of vaccine to full immunization were collected.

ADE/VED risk monitoring

After vaccination (at least 1 dose of trial vaccine) (at each visit), subjects will be reminded to contact the investigator in case of fever and/or respiratory symptoms (e.g., dyspnea, sore throat, etc.), suspected or confirmed cases of COVID-19 occurring during the study period. If the subjects are suspected or confirmed to be infected with SARS-COV-2 during the trial period, they should go to a local designated hospital for diagnosis and treatment. A detailed case-by-case investigation is required for confirmed cases. In the event of severe COVID-19 infection or death, an expert meeting should be held to evaluate ADE/VED.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 and above with full capacity for civil conduct, who can provide valid identification;
2. The subjects voluntarily agree to participate in the study and sign the informed consent to understand and comply with the requirements of the study protocol;
3. Fertile men and women of reproductive age did not have sex from day 1 of the last menstrual cycle to day 1 of the study, or did not have sex using effective contraceptive methods and did not experience contraceptive failure (examples of contraceptive failure include male condom rupture during sex). At the same time, subjects agreed to take effective contraceptive measures for 1 month from the signing of informed consent to the full immunization and no pregnancy plans during this period.

Exclusion Criteria:

1. History of novel coronavirus infection confirmed or asymptomatic infected persons or positive nucleic acid test of novel Coronavirus;
2. SARS virus history;
3. For those with fever, axillary temperature ≥37.3℃ on the day of inclusion;
4. A past history of severe allergy to any vaccine, or to the active ingredient of the test vaccine, any inactive ingredient, or substance used in the manufacturing process, including aluminum preparations, egg protein, neomycin, formaldehyde, tritonX-100, such as: Acute anaphylaxis, dyspnea, angioneurotic edema, etc., or allergies during previous vaccinations of the same kind;
5. Patients with uncontrolled epilepsy and other serious neurological diseases (e.g., transverse myelitis, Guillain-Barre syndrome, demyelinating disease, etc.);
6. Patients with acute diseases, or acute episodes of chronic diseases, or uncontrolled severe chronic diseases (such as hypertension that cannot be controlled by drugs, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg);
7. Patients at the active stage of autoimmune diseases (systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, sjogren's syndrome, etc.), patients with congenital or acquired immune deficiency, HIV infection with opportunistic infection or uncontrolled malignant tumor, lymphoma and leukemia;
8. No spleen, or splenic operation history;
9. Received immunomodulators within 6 months, such as immunosuppressive doses of glucocorticoids (dose reference: equivalent to prednisone 20mg/ day, over a week); Or monoclonal antibodies; Or thymosin; Or interferon; However, topical use (such as ointments, eye drops, inhalants or nasal sprays) is allowed;
10. Has received blood or blood-related products, including immunoglobulin (including rabies immunoglobulin and tetanus immunoglobulin), within 3 months prior to experimental vaccine vaccination; Or planned use of the experimental vaccine within 1 month of vaccination;
11. If subunit vaccine and inactivated vaccine are administered within 7 days prior to experimental vaccine inoculation, live attenuated vaccine shall be administered within 14 days prior to experimental vaccine inoculation;
12. Lactating women or pregnant women (including women of childbearing age with positive urine pregnancy test);
13. Those who have participated in or are participating in clinical trials related to COVID-19, or are participating in clinical trials of other drugs, or have received COVID-19 vaccines; The Investigator believes that the subject has any disease or condition that may place the subject at unacceptable risk; Subjects cannot meet the requirements of the program; Conditions that interfere with the assessment of vaccine response.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: | 14 days after vaccination
  Positive conversion rate of SARS-COV-2 neutralizing antibody at day 14 after full inoculation of recombinant Novel Coronavirus vaccine (CHO cells).

SECONDARY OUTCOMES:
Secondary endpoint: | 14 days after vaccination
  SARS-cov-2 neutralizing antibody GMT on day 14 after full immunization with recombinant Novel Coronavirus vaccine (CHO cells);
Secondary endpoint: | 1 months after full vaccination
  HI antibody GMT, positive conversion rate and serum protection rate of influenza virus typing 30 days after influenza vaccination;
Secondary endpoint: | 1 months after full vaccination
  Incidence of adverse reactions/events at each time point after each dose of recombinant Novel Coronavirus vaccine (CHO cells) (at least 30 min, 0-7 days and 8-30 days after inoculation);
Secondary endpoint: | within 30 minutes of influenza vaccination
  Incidence of adverse reactions/events within 30 minutes of influenza vaccination;
Secondary endpoint: | 1 months after full vaccination
  Incidence of all serious adverse events (SAE) and incidence of vaccine-related SAE from the first dose of recombinant Novel Coronavirus vaccine (CHO cells) to 1 month after full vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No